CLINICAL TRIAL: NCT07300878
Title: Comparison Of Hemodynamic Stress Response To Laryngoscopy With Video Laryngoscopy Versus Macintosh Laryngoscopy In Patients Undergoing Elective Surgeries Under General Anesthesia
Brief Title: Effect of Video Laryngoscopy Versus Conventional Laryngoscopy Upon Hemodynamics
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Muhammad Haroon Anwar, Principal Investigator, Pakistan Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F.5.2/2024(ERRC)/PIMS
Record Dates: First submitted 2025-12-21; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Laryngoscopic Stress Response; Video Laryngoscopy; Conventional Laryngoscopy
Keywords: Laryngoscopic stress response; Video laryngoscopy; Conventional laryngoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Video laryngoscopy (Experimental): Patient in this group will be intubated using hyperangulated C MAC video laryngoscope
  Interventions: Device: C MAC hyperangulated video laryngoscopy
- Conventional Laryngoscopy (Active Comparator): Patient in this group will be intubated using conventional macintosh laryngoscopic blade
  Interventions: Device: Conventional macintosh laryngoscopy

INTERVENTIONS:
Device: C MAC hyperangulated video laryngoscopy — Patient will be intubated using hyperangulated C MAC video laryngoscope
  Arms: Video laryngoscopy
Device: Conventional macintosh laryngoscopy — Patient in this group will be intubated using conventional macintosh laryngoscopy
  Arms: Conventional Laryngoscopy

SUMMARY:
In general anestheisa airway is secured by passing a tube down the widpipe. This helps the patient to breath via ventilator during anesthesia. For placing this tube laryngoscopy is done which results in increase in blood pressure and heart rate. This study will compare the rise in blood pressure and heart rate among when using video laryngoscope with conventional laryngoscope.

DETAILED DESCRIPTION:
In this study Patients will be randomly divided into two groups with group V patients being intubated using Videolaryngoscope while group M patients will be intubated using Macintosh laryngoscope. The amount of rise in blood pressure and heart rate as a result of laryngoscopy will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgeries under General Endotracheal Anesthesia. ASA class I and II.

Exclusion Criteria:

* Pregnancy

  * Body mass index >35 kg/m2
  * No teeth
  * Maxillofacial trauma
  * Limited Cervical spine movement
  * Upper Airway Tumors
  * Preoperative assessment indicating difficult airway requiring use of video laryngoscope or fiberoptic intubation.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | Upon arrival in OR (baseline) then immediately following intubation (T1) and then at 3,5,10 minutes following intubation

SECONDARY OUTCOMES:
Mean Blood Pressure | This will be measured upon arrival in OR (baseline) immediately following intubation(T1) and then at 3,5,10 minutes following intubation
Systolic Blood Pressure | This will be measured upon arrival in OR (baseline) immediately following intubation(T1) and then at 3,5,10 minutes following intubation
Diastolic Blood Pressure | This will be measured upon arrival in OR (baseline) immediately following intubation(T1) and then at 3,5,10 minutes following intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Anesthesia PIMS, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No
This is due to hospital and ethical committee policies

REFERENCES:
- [Background] Wang L, Li H, Zhong Y, Ye S, Deng J, Pan T, Zhang Y. Comparative Analysis of Hemodynamic Responses and Oropharyngeal Complications in Tracheal Intubation: Evaluating Conventional, Video, and Rigid Video Laryngoscopes Under General Anesthesia. Med Sci Monit. 2024 Sep 5;30:e944916. doi: 10.12659/MSM.944916. PMID 39233395